CLINICAL TRIAL: NCT03176446
Title: Pain and Anxiety Evaluation in Children Using Different Techniques of Local Anesthesia for Dental Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Ponta Grossa (Other)
Responsible Party: Principal Investigator, Priscila de Camargo Smolarek, PhD student, Universidade Estadual de Ponta Grossa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 64773417.3.0000.5689
Record Dates: First submitted 2017-05-12; First posted 2017-06-05 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Pediatric Dentistry; Local Anesthesia; Pain Management
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, Local; Anesthesia; Anesthetics, Local; Anesthetics

STUDY DESIGN:
Intervention Model Description: The total sample is divided into two subgroups, with 105 children aged 5 to 8 years and 105 children aged 9 to 12 years. The analysis is more sensitive and specific to each subgroup. The results of each subgroup will be analyzed in isolation and give rise to two different papers.
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Active Comparator): The children anesthesia will be traditional technique
  Interventions: Device: Local anesthesia with traditional technique; Drug: Topic anesthesia; Drug: Local anesthetic
- Computerized Group (Active Comparator): The children anesthesia will be computerized technique
  Interventions: Device: Local anesthesia with computerized technique; Drug: Topic anesthesia; Drug: Local anesthetic
- DentalVibe Group (Active Comparator): The children anesthesia will be DentalVibe technique
  Interventions: Device: Local anesthesia with DentalVibe technique; Drug: Topic anesthesia; Drug: Local anesthetic

INTERVENTIONS:
Device: Local anesthesia with traditional technique — Puncture with short needle in the region of the apical third of the tooth to be anesthetized Injection of local anesthetic, with speed 1ml / min
  Other Names: Traditional anesthesia; Conventional anesthesia
  Arms: Control Group
Device: Local anesthesia with computerized technique — Puncture with short needle in the region of the apical third of the tooth to be anesthetized according to the recommendations of the manufacturer Injection of local anesthetic with computerized anesthesia equipment, with speed 0.5 ml / min
  Other Names: Computerized anesthesia
  Arms: Computerized Group
Device: Local anesthesia with DentalVibe technique — Use of DentalVibe in the apical region of the tooth to be anesthetized according to the manufacturer's guidelines Puncture with short needle enters the tips of the DentalVibe Injection of local anesthetic with traditional carpule, with speed 1 ml / min
  Other Names: DentalVibe anesthesia
  Arms: DentalVibe Group
Drug: Topic anesthesia — Application of topical anesthetic for 60 seconds with benzocaine
  Other Names: Topical anesthesia
Drug: Local anesthetic — 2% lidocaine with epinephrine 1: 100000 1.8 mL
  Other Names: Anesthetic

SUMMARY:
Fear and dental anxiety are often associated with the use of needles and syringes for local anesthesia, and painful perception during the administration of local anesthetics is often the main reason for anxiety behaviors and defensive reactions. Dental trauma originates in childhood, through experience misconduct. The objective of this study is to evaluate the pain and anxiety related to 4 different modalities of anesthesia in children. Will be selected volunteers aged between 5 and 12 years who need restorative dental treatment in posterior teeth in the upper 2 quadrants. All patients will receive 1 modality of anesthesia: conventional anesthesia (control group), computerized anesthesia, Dental Vibe anesthesia and computerized anesthesia + DentalVibe anesthesia. Evaluations will be made with physiological and behavioral criteria. For the physiological evaluation will be measured the blood pressure, respiratory rate, heart rate, oximetry and salivary cortisol before and during each anesthesia. As criteria for evaluation of anxiety will be applied the methods, Corah and modified VPT before anesthesia and modified VPT will be repeated after anesthesia. The pain will be assessed at the end of each anesthesia with Visual Analogue Scale (VAS) and Wong Baker Faces. The results will be submitted to parametric and non-parametric statistical analysis, according to the data obtained in the different evaluation criteria.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes, aged between 5 and 12 years, requiring dental treatment under local anesthesia in the first permanent molars or deciduous maxilla.

Exclusion Criteria:

* The person responsible does not authorize the participation of the child as a research volunteer.
* Be using pain modulating drugs.
* Be using anxiety modulating drugs.
* Patients with a history of hypersensitivity to local anesthetics.
* Patients with a history of systemic diseases.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Self-perception of pain | Immediately after anesthesia
  The pain will be analyzed by the Wong Baker Faces scales
Pain Behavior | During the anesthetic procedure
  The pain will be analyzed by the FLACC
Self-perception of pain | Immediately after anesthesia
  The pain will be analyzed by the Visual Analogue Scale (0-10). 0- no pain, 10- severe pain

SECONDARY OUTCOMES:
SCARED Questionnaire | Before anesthesia
  Children will be evaluated for the anxiety behavior prior to any anesthesia by answering the SCARED questionnaire
Corah Questionnaire | Before anethesia
  Children will be evaluated for the dentistry anxiety prior to any anesthesia
VPT modified | Before anethesia and immediately after anesthesia
  Children will be evaluated for the anxiety after to any anesthesia
Blood pressure | Immediately before anesthesia, during anesthesia
  The physiological response of anxiety to local dental anesthesia will be evaluated by parameters of blood pressure
Respiratory rate | Immediately before anesthesia, during anesthesia
  The physiological response of anxiety to local dental anesthesia will be evaluated by parameters of respiratory rate
Heart rate | Immediately before anesthesia, during anesthesia
  The physiological response of anxiety to local dental anesthesia will be evaluated by parameters of heart rate
Oxygen saturation | Immediately before anesthesia, during anesthesia
  The physiological response of anxiety to local dental anesthesia will be evaluated by parameters of oxygen saturation
Salivary cortisol | Immediately before anesthesia, during anesthesia
  The physiological response of anxiety to local dental anesthesia will be evaluated by parameters of salivary cortisol

CONTACTS AND LOCATIONS:
Locations (1):
- Ponta Grossa State University, Ponta Grossa, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Approval of the ethics committee: 1.941.369 — http://plataformabrasil.saude.gov.br